CLINICAL TRIAL: NCT01644734
Title: MATHS: Assessment of Health-status of Patients With COPD on MAintenance THerapy With Spiriva® HH Measured by CAT Test
Brief Title: Assessment of Health-status of Patients With Chronic Obstructive Pulmonary Disease (COPD) on Maintenance Therapy With Spiriva HH Measured by COPD Assessment Test (CAT) Test
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group
Other Study IDs: 205.502
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Drug: Spiriva HandiHaler

SUMMARY:
To evaluate the early (3-month) impact of the long-acting anticholinergic Spiriva HH maintenance treatment on the COPD symptoms using the novel COPD Assessment test (CAT) in the real life setting of COPD patients, previously treated with short-acting bronchodilator on regular or as-needed basis.

ELIGIBILITY:
Inclusion criteria:

* Male and female ambulatory outpatients being seen in a participating physicians office for routine care,
* Patients with a clinical diagnosis of COPD (all stages according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines 2010) being treated with long-acting anticholinergic (Tiotropium, Spiriva® HandiHaler® ) as maintenance therapy within the product label and a maximum of the last 4 weeks (0.-28. days before Visit 1),
* Patients previously treated with short-acting bronchodilators on regular or as-needed basis for at least 3 months before change to long-acting anticholinergic treatment,
* Patient fluent in language of questionnaire and having the cognitive and functional abilities required to fill in the questionnaire alone.

Exclusion criteria:

* Uncooperative patients as judged by the physician,
* Patients with any conditions excluded as per Country specific package insert,
* Patients currently enrolled in any clinical trial,
* Patients with COPD exacerbation or any acute disease in the last 3 months before Visit 1.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1328 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (247):
- Poland (247):
  - Boehringer Ingelheim Investigational Site 236, Andrychów
  - Boehringer Ingelheim Investigational Site 170, Bialystok
  - Boehringer Ingelheim Investigational Site 184, Bialystok
  - Boehringer Ingelheim Investigational Site 240, Bialystok
  - Boehringer Ingelheim Investigational Site 44, Bialystok
  - Boehringer Ingelheim Investigational Site 84, Bialystok
  - Boehringer Ingelheim Investigational Site 33, Bielsko-Biala
  - Boehringer Ingelheim Investigational Site 34, Bielsko-Biala
  - Boehringer Ingelheim Investigational Site 35, Bielsko-Biala
  - Boehringer Ingelheim Investigational Site 79, Biskupiec
  - Boehringer Ingelheim Investigational Site 116, Bochnia
  - Boehringer Ingelheim Investigational Site 115, Brzesko
  - Boehringer Ingelheim Investigational Site 138, Brzesko
  - Boehringer Ingelheim Investigational Site 185, Brzeziny
  - Boehringer Ingelheim Investigational Site 90, Brzozów
  - Boehringer Ingelheim Investigational Site 105, Bydgoszcz
  - Boehringer Ingelheim Investigational Site 119, Bydgoszcz
  - Boehringer Ingelheim Investigational Site 123, Bydgoszcz
  - Boehringer Ingelheim Investigational Site 222, Bydgoszcz
  - Boehringer Ingelheim Investigational Site 27, Bydgoszcz
  - Boehringer Ingelheim Investigational Site 21, Chełm
  - Boehringer Ingelheim Investigational Site 22, Chełm
  - Boehringer Ingelheim Investigational Site 11, Chełmsko Śląskie
  - Boehringer Ingelheim Investigational Site 233, Chodzież
  - Boehringer Ingelheim Investigational Site 226, Chojnice
  - Boehringer Ingelheim Investigational Site 149, Chorzów
  - Boehringer Ingelheim Investigational Site 153, Chorzów
  - Boehringer Ingelheim Investigational Site 88, Ciechanów
  - Boehringer Ingelheim Investigational Site 232, Czarnków
  - Boehringer Ingelheim Investigational Site 229, Częstochowa
  - Boehringer Ingelheim Investigational Site 4, Częstochowa
  - Boehringer Ingelheim Investigational Site 23, Dąbrowa Górnicza
  - Boehringer Ingelheim Investigational Site 92, Domaradz
  - Boehringer Ingelheim Investigational Site 246, Dziergowice
  - Boehringer Ingelheim Investigational Site 133, Gdansk
  - Boehringer Ingelheim Investigational Site 134, Gdansk
  - Boehringer Ingelheim Investigational Site 136, Gdansk
  - Boehringer Ingelheim Investigational Site 155, Gdansk
  - Boehringer Ingelheim Investigational Site 156, Gdansk
  - Boehringer Ingelheim Investigational Site 20, Gdansk
  - Boehringer Ingelheim Investigational Site 234, Gdansk
  - Boehringer Ingelheim Investigational Site 31, Gdansk
  - Boehringer Ingelheim Investigational Site 41, Gdynia
  - Boehringer Ingelheim Investigational Site 217, Gliwice
  - Boehringer Ingelheim Investigational Site 243, Gmina Jędrzejów
  - Boehringer Ingelheim Investigational Site 141, Gmina Końskie
  - Boehringer Ingelheim Investigational Site 142, Gmina Końskie
  - Boehringer Ingelheim Investigational Site 73, Gmina Sawin
  - Boehringer Ingelheim Investigational Site 107, Gmina Śrem
  - Boehringer Ingelheim Investigational Site 213, Gmina Śrem
  - Boehringer Ingelheim Investigational Site 181, Gmina Świecie
  - Boehringer Ingelheim Investigational Site 38, Gmina Uchanie
  - Boehringer Ingelheim Investigational Site 50, Gorzów Wielkopolski
  - Boehringer Ingelheim Investigational Site 85, Góra
  - Boehringer Ingelheim Investigational Site 174, Grodzisk Mazowiecki
  - Boehringer Ingelheim Investigational Site 176, Grodzisk Mazowiecki
  - Boehringer Ingelheim Investigational Site 56, Gryfice
  - Boehringer Ingelheim Investigational Site 247, Głuchołazy
  - Boehringer Ingelheim Investigational Site 179, Jarosław
  - Boehringer Ingelheim Investigational Site 108, Jasło
  - Boehringer Ingelheim Investigational Site 225, Jasło
  - Boehringer Ingelheim Investigational Site 8, Jasło
  - Boehringer Ingelheim Investigational Site 148, Jelenia Góra
  - Boehringer Ingelheim Investigational Site 162, Katowice
  - Boehringer Ingelheim Investigational Site 163, Katowice
  - Boehringer Ingelheim Investigational Site 164, Katowice
  - Boehringer Ingelheim Investigational Site 212, Katowice
  - Boehringer Ingelheim Investigational Site 69, Kcynia
  - Boehringer Ingelheim Investigational Site 112, Kielce
  - Boehringer Ingelheim Investigational Site 18, Kielce
  - Boehringer Ingelheim Investigational Site 19, Kielce
  - Boehringer Ingelheim Investigational Site 219, Konin
  - Boehringer Ingelheim Investigational Site 51, Koszalin
  - Boehringer Ingelheim Investigational Site 52, Koszalin
  - Boehringer Ingelheim Investigational Site 49, Kołobrzeg
  - Boehringer Ingelheim Investigational Site 122, Krakow
  - Boehringer Ingelheim Investigational Site 135, Krakow
  - Boehringer Ingelheim Investigational Site 143, Krakow
  - Boehringer Ingelheim Investigational Site 146, Krakow
  - Boehringer Ingelheim Investigational Site 171, Krakow
  - Boehringer Ingelheim Investigational Site 177, Krakow
  - Boehringer Ingelheim Investigational Site 214, Krakow
  - Boehringer Ingelheim Investigational Site 87, Krakow
  - Boehringer Ingelheim Investigational Site 94, Krakow
  - Boehringer Ingelheim Investigational Site 129, Kraśnik
  - Boehringer Ingelheim Investigational Site 204, Kraśnik
  - Boehringer Ingelheim Investigational Site 207, Kraśnik
  - Boehringer Ingelheim Investigational Site 192, Krosno
  - Boehringer Ingelheim Investigational Site 194, Kutno
  - Boehringer Ingelheim Investigational Site 13, Kłodzko
  - Boehringer Ingelheim Investigational Site 97, Legionowo
  - Boehringer Ingelheim Investigational Site 86, Lędziny
  - Boehringer Ingelheim Investigational Site 127, Liśnik Duży
  - Boehringer Ingelheim Investigational Site 187, Lodz
  - Boehringer Ingelheim Investigational Site 188, Lodz
  - Boehringer Ingelheim Investigational Site 193, Lodz
  - Boehringer Ingelheim Investigational Site 198, Lodz
  - Boehringer Ingelheim Investigational Site 206, Lodz
  - Boehringer Ingelheim Investigational Site 186, Lowicz
  - Boehringer Ingelheim Investigational Site 158, Lubań
  - Boehringer Ingelheim Investigational Site 37, Lubartów
  - Boehringer Ingelheim Investigational Site 172, Lubin
  - Boehringer Ingelheim Investigational Site 173, Lubin
  - Boehringer Ingelheim Investigational Site 196, Lubin
  - Boehringer Ingelheim Investigational Site 124, Lublin
  - Boehringer Ingelheim Investigational Site 17, Lublin
  - Boehringer Ingelheim Investigational Site 29, Lublin
  - Boehringer Ingelheim Investigational Site 7, Lublin
  - Boehringer Ingelheim Investigational Site 242, Lubliniec
  - Boehringer Ingelheim Investigational Site 209, Luboń
  - Boehringer Ingelheim Investigational Site 106, Ludwikowo
  - Boehringer Ingelheim Investigational Site 45, Maków Mazowiecki
  - Boehringer Ingelheim Investigational Site 168, Malbork
  - Boehringer Ingelheim Investigational Site 110, Mielec
  - Boehringer Ingelheim Investigational Site 159, Milicz
  - Boehringer Ingelheim Investigational Site 25, Myszków
  - Boehringer Ingelheim Investigational Site 150, Mysłowice
  - Boehringer Ingelheim Investigational Site 215, Nisko
  - Boehringer Ingelheim Investigational Site 128, Nowy Dwór Gdański
  - Boehringer Ingelheim Investigational Site 109, Nowy Sącz
  - Boehringer Ingelheim Investigational Site 72, Olecko
  - Boehringer Ingelheim Investigational Site 36, Olsztyn
  - Boehringer Ingelheim Investigational Site 245, Opatów
  - Boehringer Ingelheim Investigational Site 114, Ostrowiec Świętokrzyski
  - Boehringer Ingelheim Investigational Site 145, Ostrowiec Świętokrzyski
  - Boehringer Ingelheim Investigational Site 154, Oława
  - Boehringer Ingelheim Investigational Site 237, Pabianice
  - Boehringer Ingelheim Investigational Site 182, Papowo Biskupie
  - Boehringer Ingelheim Investigational Site 216, Pawonków
  - Boehringer Ingelheim Investigational Site 189, Piekary Śląskie
  - Boehringer Ingelheim Investigational Site 32, Pietrzykowice
  - Boehringer Ingelheim Investigational Site 203, Piotrkow Trybunalski
  - Boehringer Ingelheim Investigational Site 40, Piła
  - Boehringer Ingelheim Investigational Site 93, Pniewy
  - Boehringer Ingelheim Investigational Site 130, Poniatowa
  - Boehringer Ingelheim Investigational Site 201, Poznan
  - Boehringer Ingelheim Investigational Site 208, Poznan
  - Boehringer Ingelheim Investigational Site 227, Poznan
  - Boehringer Ingelheim Investigational Site 228, Poznan
  - Boehringer Ingelheim Investigational Site 231, Poznan
  - Boehringer Ingelheim Investigational Site 126, Prabuty
  - Boehringer Ingelheim Investigational Site 218, Proszowice
  - Boehringer Ingelheim Investigational Site 131, Pruszcz Gdański
  - Boehringer Ingelheim Investigational Site 191, Przemyśl
  - Boehringer Ingelheim Investigational Site 59, Płock
  - Boehringer Ingelheim Investigational Site 169, Rabka-Zdrój
  - Boehringer Ingelheim Investigational Site 117, Radom
  - Boehringer Ingelheim Investigational Site 118, Radom
  - Boehringer Ingelheim Investigational Site 151, Ruda Śląska
  - Boehringer Ingelheim Investigational Site 152, Ruda Śląska
  - Boehringer Ingelheim Investigational Site 230, Ruda Śląska
  - Boehringer Ingelheim Investigational Site 82, Ruda Śląska
  - Boehringer Ingelheim Investigational Site 180, Rumia
  - Boehringer Ingelheim Investigational Site 239, Rumia
  - Boehringer Ingelheim Investigational Site 5, Rumia
  - Boehringer Ingelheim Investigational Site 104, Rybnik
  - Boehringer Ingelheim Investigational Site 183, Rybnik
  - Boehringer Ingelheim Investigational Site 83, Rybnik
  - Boehringer Ingelheim Investigational Site 175, Rzeszów
  - Boehringer Ingelheim Investigational Site 178, Rzeszów
  - Boehringer Ingelheim Investigational Site 190, Sanok
  - Boehringer Ingelheim Investigational Site 78, Sejny
  - Boehringer Ingelheim Investigational Site 160, Siewierz
  - Boehringer Ingelheim Investigational Site 241, Skarżysko-Kamienna
  - Boehringer Ingelheim Investigational Site 157, Skawina
  - Boehringer Ingelheim Investigational Site 10, Skoczów
  - Boehringer Ingelheim Investigational Site 167, Skrzyszów
  - Boehringer Ingelheim Investigational Site 14, Sokołowsko
  - Boehringer Ingelheim Investigational Site 113, Sopot
  - Boehringer Ingelheim Investigational Site 166, Sosnowiec
  - Boehringer Ingelheim Investigational Site 24, Sosnowiec
  - Boehringer Ingelheim Investigational Site 125, Stalowa Wola
  - Boehringer Ingelheim Investigational Site 144, Starachowice
  - Boehringer Ingelheim Investigational Site 80, Starachowice
  - Boehringer Ingelheim Investigational Site 120, Stargard
  - Boehringer Ingelheim Investigational Site 95, Sucha Beskidzka
  - Boehringer Ingelheim Investigational Site 16, Supraśl
  - Boehringer Ingelheim Investigational Site 54, Suwałki
  - Boehringer Ingelheim Investigational Site 55, Suwałki
  - Boehringer Ingelheim Investigational Site 76, Syców
  - Boehringer Ingelheim Investigational Site 43, Szczecin
  - Boehringer Ingelheim Investigational Site 48, Szczecin
  - Boehringer Ingelheim Investigational Site 61, Szczecin
  - Boehringer Ingelheim Investigational Site 66, Szczecin
  - Boehringer Ingelheim Investigational Site 67, Szczecin
  - Boehringer Ingelheim Investigational Site 26, Szczecinek
  - Boehringer Ingelheim Investigational Site 53, Sławno
  - Boehringer Ingelheim Investigational Site 96, Słubice
  - Boehringer Ingelheim Investigational Site 205, Słupca
  - Boehringer Ingelheim Investigational Site 1, Świdnik
  - Boehringer Ingelheim Investigational Site 111, Tarnobrzeg
  - Boehringer Ingelheim Investigational Site 224, Tarnobrzeg
  - Boehringer Ingelheim Investigational Site 200, Tarnowskie Góry
  - Boehringer Ingelheim Investigational Site 139, Tarnów
  - Boehringer Ingelheim Investigational Site 140, Tarnów
  - Boehringer Ingelheim Investigational Site 101, Torun
  - Boehringer Ingelheim Investigational Site 70, Torun
  - Boehringer Ingelheim Investigational Site 71, Torun
  - Boehringer Ingelheim Investigational Site 220, Trzcianka Lubuska
  - Boehringer Ingelheim Investigational Site 103, Twardogóra
  - Boehringer Ingelheim Investigational Site 147, Tychy
  - Boehringer Ingelheim Investigational Site 244, Tychy
  - Boehringer Ingelheim Investigational Site 100, Warsaw
  - Boehringer Ingelheim Investigational Site 121, Warsaw
  - Boehringer Ingelheim Investigational Site 137, Warsaw
  - Boehringer Ingelheim Investigational Site 161, Warsaw
  - Boehringer Ingelheim Investigational Site 165, Warsaw
  - Boehringer Ingelheim Investigational Site 210, Warsaw
  - Boehringer Ingelheim Investigational Site 223, Warsaw
  - Boehringer Ingelheim Investigational Site 238, Warsaw
  - Boehringer Ingelheim Investigational Site 2, Warsaw
  - Boehringer Ingelheim Investigational Site 3, Warsaw
  - Boehringer Ingelheim Investigational Site 42, Warsaw
  - Boehringer Ingelheim Investigational Site 46, Warsaw
  - Boehringer Ingelheim Investigational Site 74, Warsaw
  - Boehringer Ingelheim Investigational Site 91, Warsaw
  - Boehringer Ingelheim Investigational Site 99, Warsaw
  - Boehringer Ingelheim Investigational Site 39, Wałcz
  - Boehringer Ingelheim Investigational Site 6, Wejherowo
  - Boehringer Ingelheim Investigational Site 199, Wieliczna
  - Boehringer Ingelheim Investigational Site 235, Wieluń
  - Boehringer Ingelheim Investigational Site 197, Witonia
  - Boehringer Ingelheim Investigational Site 65, Wloc³awek
  - Boehringer Ingelheim Investigational Site 28, Wodzisław Śląski
  - Boehringer Ingelheim Investigational Site 98, Wołomin
  - Boehringer Ingelheim Investigational Site 102, Wroclaw
  - Boehringer Ingelheim Investigational Site 202, Wroclaw
  - Boehringer Ingelheim Investigational Site 221, Wroclaw
  - Boehringer Ingelheim Investigational Site 62, Wroclaw
  - Boehringer Ingelheim Investigational Site 63, Wroclaw
  - Boehringer Ingelheim Investigational Site 64, Wroclaw
  - Boehringer Ingelheim Investigational Site 89, Wroclaw
  - Boehringer Ingelheim Investigational Site 68, Zabrze
  - Boehringer Ingelheim Investigational Site 75, Zabrze
  - Boehringer Ingelheim Investigational Site 77, Zabrze
  - Boehringer Ingelheim Investigational Site 12, Ząbkowice Śląskie
  - Boehringer Ingelheim Investigational Site 9, Ząbkowice Śląskie
  - Boehringer Ingelheim Investigational Site 60, Zągoty
  - Boehringer Ingelheim Investigational Site 132, Zblewo
  - Boehringer Ingelheim Investigational Site 195, Zgierz
  - Boehringer Ingelheim Investigational Site 15, Zielona Góra
  - Boehringer Ingelheim Investigational Site 47, Zielona Góra
  - Boehringer Ingelheim Investigational Site 81, Zielonka k/Warszawy
  - Boehringer Ingelheim Investigational Site 211, Żyrardów
  - Boehringer Ingelheim Investigational Site 57, Łomża
  - Boehringer Ingelheim Investigational Site 58, Łomża
  - Boehringer Ingelheim Investigational Site 30, Łuków

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 46 patients were not documented to be treated with the study drug.
Groups:
- Patients Treated With Spiriva HandiHaler: Inhalator is administered once daily in the dosage of 18µg.
Period: Overall Study
Arm/Group | Patients Treated With Spiriva HandiHaler
Started | 1282 (Patients with documentation of treatment.)
Completed | 1016
Not Completed | 266
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 17
Not completed — Reasons other than stated above | 7
Not completed — Missing documentation | 238

BASELINE CHARACTERISTICS:
Population: Patients from the Treated Set (TS) which are dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Arm/Group | Patients Treated With Spiriva HandiHaler
Number analyzed (Participants) | 1282
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 494
  Male | 788

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Maintaining or Improving Their Health Status
Description: The health status was measured by the total COPD Assessment Test (CAT) score at baseline and at the end of the observation period after app. 3 months (visit 3). Therefore, the total CAT score at baseline and at Visit 3 was calculated by adding up the scores of the single questions of the CAT questionnaire. In the case of one or more missing items the total score was not determined for the specific visit. The health status is considered to be maintained or improved if the change in the total CAT score from baseline at Visit 3 is ≥0.
Time Frame: Baseline, 3 months
Population: Patients from the Full Analysis Set (FAS) which includes all patients in the treated set and who have valid CAT questionnaire results both at baseline and at visit 3.
Measure: Number; unit: participants
Arm/Group | Patients Treated With Spiriva HandiHaler
Number analyzed (Participants) | 1016
participants | 972 [94.2 to 96.8]

2. Secondary Outcome: Change in the Total CAT Score (Value Baseline Minus 3 Months)
Description: The change represents the value at baseline minus the value after 3 months. The total CAT score ranges from 0 to 40 where 0 represents no symptoms and 40 very bad symptoms. Therefore, a positive value for the change in the total CAT score means an improvement.
Time Frame: Baseline, 3 months
Population: Patients from FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Treated With Spiriva HandiHaler
Number analyzed (Participants) | 1016
units on a scale | 7.0 (5.9)
Statistical Analysis 1: Comparison: Patients Treated With Spiriva HandiHaler; Null hypothesis: no change in the total CAT score between baseline and after 3 months; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Average of 92.4 days
Arm/Group | Patients Treated With Spiriva HandiHaler
Serious Adverse Events (participants affected / at risk) | 0/1282
Other Adverse Events (participants affected / at risk) | 0/1282

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.